CLINICAL TRIAL: NCT07206732
Title: Ultrasound-Guided Inferior Vena Cava Assessment Versus Central Venous Pressure Monitoring in Early and Post-Resuscitation Detection of Hypovolemia Among Shocked Patients in the Emergency Department
Brief Title: IVC Ultrasound Versus Central Venous Pressure for Early Detection of Hypovolemia in Shock Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mohamed Abd Elgwad, Principal Investigator at Emergency Medicine department Assiut University, Assiut University
Other Study IDs: IVC-CVP-ShockED-2025
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Shock; Hypovolemia; Circulatory Failure
Keywords: Shock; Hypovolemia; Emergency department; Central venous pressure; Fliud resuscitation; Ultrasound guided IVC
MeSH Terms: conditions — Shock; Hypovolemia; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound-Guided Inferior Vena Cava Assessment — This intervention involves bedside ultrasound measurement of the inferior vena cava (IVC) diameter and calculation of the IVC collapsibility/distensibility index. Assessments will be performed both at initial presentation and after fluid resuscitation in shock patients. The procedure is non-invasive, rapid, and performed according to standardized emergency ultrasound protocols, distinguishing it from invasive monitoring methods.

SUMMARY:
This study aims to compare ultrasound-guided inferior vena cava (IVC) assessment with central venous pressure (CVP) monitoring for the detection of hypovolemia in shock patients in the emergency department. The primary objective is to evaluate the diagnostic accuracy and clinical utility of IVC collapsibility index compared to CVP values in both early and post-resuscitation phases. The study will prospectively enroll shock patients, collect demographic and clinical data, and analyze the correlation between IVC and CVP measurements to determine their role in guiding fluid resuscitation and hemodynamic management.

DETAILED DESCRIPTION:
Hypovolemia is a major contributor to morbidity and mortality among patients presenting with shock in the emergency department. Early recognition and accurate assessment of intravascular volume status are essential for effective resuscitation. Central venous pressure (CVP) monitoring has traditionally been used but is invasive and may not always accurately reflect volume status. Ultrasound-guided inferior vena cava (IVC) assessment offers a non-invasive alternative, with the IVC collapsibility index shown to correlate with volume responsiveness. This prospective observational study will enroll patients diagnosed with shock and compare IVC measurements with CVP values during both early presentation and post-resuscitation phases. The findings are expected to provide evidence on the diagnostic agreement between IVC ultrasound and CVP monitoring, potentially supporting the use of IVC ultrasound as a rapid, reliable, and less invasive tool for guiding fluid therapy in emergency settings.

ELIGIBILITY:
Inclusion Criteria:

1- Adult patients aged ≥18 years. 2.Both male and female patients will be included in the study. 3. Presentation to the Emergency Department with clinical evidence of shock, defined by: Hypotension (systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg).

Evidence of tissue hypoperfusion (e.g., altered mental status, cold extremities, or oliguria).

Elevated serum lactate (>2 mmol/L). 4. Shock attributed to hypovolemic, septic, or hemorrhagic etiologies. 5. Patients requiring fluid resuscitation and hemodynamic monitoring.

Exclusion Criteria:

1 - Patients younger than 18 years. 2. Pregnancy. 3.Cardiogenic or obstructive shock (e.g., cardiac tamponade, massive pulmonary embolism, or tension pneumothorax).

4.Known inferior vena cava (IVC) anomalies (e.g., congenital absence, thrombosis).

5. Increased intra-abdominal pressure or severe ascites. 6. Morbid obesity (BMI ≥40 kg/m²) or any condition interfering with adequate IVC ultrasound visualization.

7. Prior central venous catheterization performed before Emergency Department arrival.

8. Congestive heart failure (CHF) with left ventricular ejection fraction (LVEF <40%) or pulmonary hypertension.

9. Refusal of the patient or legal guardian to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients aged 18-65 years presenting with shock to the emergency department and requiring volume status assessment through both IVC ultrasound and central venous pressure monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Correlation Between IVC Collapsibility Index and Central Venous Pressure | IVC assessment will be performed at presentation and 1 hour post-resuscitation, while CVP will be monitored continuously during the first 6 hours after ED admission.
  The primary outcome is to assess the diagnostic agreement between ultrasound-guided inferior vena cava (IVC) collapsibility index and central venous pressure (CVP) values in detecting hypovolemia among shock patients in the emergency department. Measurements will be collected at two time points: during early presentation and after initial fluid resuscitation. The outcome will be evaluated by analyzing correlation coefficients, sensitivity, and specificity of IVC measurements compared with CVP

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Attia, Professor of Anathesia and ICU, Principal Investigator — Assit University; Ahmed M Mandor, Consultant of Anathesia ICU, Study Director — Assiut University; Walaa M Adel, Lecture of emergency medicine, Study Director — Seuz canal University
Locations (1):
- Emeregency medicine department ,Assiut University, Asyut, Sahel Selim, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is conducted as part of an academic thesis project. Data are limited to internal use within the research team and protected by institutional and ethical regulations.